CLINICAL TRIAL: NCT03141177
Title: A Phase 3, Randomized, Open-Label Study of Nivolumab Combined With Cabozantinib Versus Sunitinib in Participants With Previously Untreated Advanced or Metastatic Renal Cell Carcinoma
Brief Title: A Study of Nivolumab Combined With Cabozantinib Compared to Sunitinib in Previously Untreated Advanced or Metastatic Renal Cell Carcinoma
Acronym: CheckMate 9ER
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Exelixis (Industry); Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-9ER; 2017-000759-20 (EudraCT Number)
Record Dates: First submitted 2017-05-03; First posted 2017-05-04 (Actual); Results first posted 2022-04-26 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-05

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Nivolumab; cabozantinib; Sunitinib; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Doublet (Experimental): Nivolumab and Cabozantinib
  Interventions: Biological: Nivolumab; Drug: Cabozantinib
- Monotherapy (Active Comparator): Sunitinib
  Interventions: Drug: Sunitinib
- Triplet (Experimental): Nivolumab, Ipilimumab, Cabozantinib
  *Enrollment to the triplet arm was discontinued by protocol amendment
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified day
  Other Names: Opdivo; BMS-936558
  Arms: Doublet
Drug: Cabozantinib — Specified dose on specified days
  Other Names: Cabometyx
  Arms: Doublet
Drug: Sunitinib — Specified dose on specified days.
  Other Names: Sutent
  Arms: Monotherapy
Biological: Ipilimumab — Specified dose on specified days
  Other Names: Yervoy; BMS-734016
  Arms: Triplet

SUMMARY:
The purpose of this study is to determine whether Nivolumab Combined with Cabozantinib is safe and effective compared to Sunitinib in previously untreated advanced or metastatic renal cell carcinoma

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histological confirmation of RCC with a clear-cell component, including participants who may also have sarcomatoid features
* Advanced (not amenable to curative surgery or radiation therapy) or metastatic (AJCC Stage IV) RCC
* No prior systemic therapy for RCC with the following exception:

  i) One prior adjuvant or neoadjuvant therapy for completely resectable RCC if such therapy did not include an agent that targets VEGF or VEGF receptors and if recurrence occurred at least 6 months after the last dose of adjuvant or neoadjuvant therapy

Exclusion Criteria:

* Any active CNS metastases
* Any active, known or suspected autoimmune disease
* Any condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization
* Participants who have received a live/attenuated vaccine within 30 days of first treatment

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 701 (Actual)
Dates: Start 2017-07-23 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2026-01-16 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (135):
- United States (30):
  - Local Institution - 0077, Daphne, Alabama
  - Local Institution - 0044, Goodyear, Arizona
  - Local Institution - 0132, Tucson, Arizona
  - Local Institution - 0133, Bakersfield, California
  - Local Institution - 0093, Los Angeles, California
  - Local Institution - 0090, Redondo Beach, California
  - Local Institution - 0088, San Luis Obispo, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Local Institution - 0103, Aurora, Colorado
  - Local Institution - 0127, Athens, Georgia
  - Local Institution - 0086, Newnan, Georgia
  - Local Institution - 0036, Chicago, Illinois
  - Local Institution - 0042, Zion, Illinois
  - Local Institution - 0091, Fort Wayne, Indiana
  - Local Institution - 0087, Wichita, Kansas
  - Local Institution - 0113, Boston, Massachusetts
  - Local Institution - 0037, Boston, Massachusetts
  - Local Institution - 0106, Kansas City, Missouri
  - Local Institution - 0035, St Louis, Missouri
  - Local Institution - 0102, Las Vegas, Nevada
  - Local Institution - 0040, Buffalo, New York
  - Local Institution - 0017, New York, New York
  - Local Institution - 0067, Portland, Oregon
  - Local Institution - 0135, Allentown, Pennsylvania
  - Local Institution - 0105, Nashville, Tennessee
  - Local Institution - 0080, Austin, Texas
  - Local Institution - 0075, Dallas, Texas
  - Local Institution - 0068, Houston, Texas
  - Local Institution - 0078, Sherman, Texas
  - Local Institution - 0131, Norfolk, Virginia
- Argentina (7):
  - Local Institution - 0046, CABA, Buenos Aires
  - Local Institution - 0048, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Local Institution - 0114, Viedma, Río Negro Province
  - Local Institution - 0138, CABA
  - Local Institution - 0050, Córdoba
  - Local Institution - 0049, Córdoba
  - Local Institution - 0047, San Miguel de Tucumán
- Australia (10):
  - Local Institution - 0002, North Ryde, New South Wales
  - Local Institution - 0008, Sydney, New South Wales
  - Local Institution - 0009, Sydney, New South Wales
  - Local Institution - 0073, Westmead, New South Wales
  - Local Institution - 0006, Herston, Queensland
  - Local Institution - 0001, Southport, Queensland
  - Local Institution - 0004, Elizabeth Vale, South Australia
  - Local Institution - 0005, Malvern, Victoria
  - Local Institution - 0007, Doubleview, Western Australia
  - Local Institution - 0129, South Brisbane
- Brazil (8):
  - Local Institution - 0057, Belo Horizonte, Minas Gerais
  - Local Institution - 0119, Ijuí, Rio Grande do Sul
  - Local Institution - 0056, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0060, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0058, Barretos, São Paulo
  - Local Institution - 0066, Rio de Janeiro
  - Local Institution - 0074, São Paulo
  - Local Institution - 0061, São Paulo
- Local Institution - 0045, Santiago, Santiago Metropolitan, Chile
- Czechia (2):
  - Local Institution - 0034, Hradec Králové
  - Local Institution - 0033, Olomouc
- Germany (7):
  - Local Institution - 0013, Aachen
  - Local Institution - 0016, Bonn
  - Local Institution - 0117, Essen
  - Local Institution - 0023, Jena
  - Local Institution - 0010, München
  - Local Institution - 0014, Nuremberg
  - Local Institution - 0011, Tübingen
- Greece (2):
  - Local Institution - 0082, Athens
  - Local Institution - 0083, Thessaloniki
- Israel (4):
  - Local Institution - 0072, Haifa
  - Local Institution - 0070, Kfar Saba
  - Local Institution - 0071, Petah Tikva
  - Local Institution - 0069, Ramat Gan
- Italy (7):
  - Local Institution - 0054, Arezzo
  - Local Institution - 0052, Milan
  - Local Institution - 0055, Napoli
  - Local Institution - 0053, Padua
  - Local Institution - 0051, Pavia
  - Local Institution - 0147, Pavia
  - Local Institution - 0172, Terni
- Japan (25):
  - Local Institution - 0148, Akita, Akita
  - Local Institution - 0156, Hirosaki, Aomori
  - Local Institution - 0164, Sapporo, Hokkaido
  - Local Institution - 0157, Sapporo, Hokkaido
  - Local Institution - 0168, Kobe, Hyōgo
  - Local Institution - 0159, Morioka, Iwate
  - Local Institution - 0171, Yokohama, Kanagawa
  - Local Institution - 0166, Yokohama, Kanagawa
  - Local Institution - 0150, Niigata, Niigata
  - Local Institution - 0169, Okayama, Okayama-ken
  - Local Institution - 0170, Osaka, Osaka
  - Local Institution - 0160, Osakasayamashi, Osaka
  - Local Institution - 0163, Suita-shi, Osaka
  - Local Institution - 0154, Osaka, Osaka-shi
  - Local Institution - 0155, Hidaka-shi, Saitama
  - Local Institution - 0153, Tokushima, Tokushima
  - Local Institution - 0152, Adachi-ku, Tokyo
  - Local Institution - 0158, Bunkyo-ku, Tokyo
  - Local Institution - 0151, Bunkyo-ku, Tokyo
  - Local Institution - 0173, Minato-ku, Tokyo
  - Local Institution - 0167, Chiba
  - Local Institution - 0161, Fukuoka
  - Local Institution - 0162, Nagasaki
  - Local Institution - 0149, Tokyo
  - Local Institution - 0165, Yamagata
- Mexico (9):
  - Local Institution - 0108, Zapopan, Jalisco
  - Local Institution - 0062, Mexico City, Mexico City
  - Local Institution - 0116, Mexico City, Mexico City
  - Local Institution - 0115, Tlalpan, Mexico City
  - Local Institution - 0065, Monterrey, Nuevo León
  - Local Institution - 0143, Monterrey, Nuevo León
  - Local Institution - 0064, Monterrey, Nuevo León
  - Local Institution - 0063, Querétaro City, Querétaro
  - Local Institution - 0136, Mérida, Yucatán
- Poland (3):
  - Local Institution - 0084, Biała Podlaska
  - Local Institution - 0130, Bydgoszcz
  - Local Institution - 0085, Gdansk
- Romania (2):
  - Local Institution - 0021, Cluj-Napoca
  - Local Institution - 0022, Craiova
- Russia (2):
  - Local Institution - 0020, Moscow
  - Local Institution - 0099, Saint Petersburg
- Spain (6):
  - Local Institution - 0125, Barcelona
  - Local Institution - 0121, Madrid
  - Local Institution - 0120, Madrid
  - Local Institution - 0144, Santander
  - Local Institution - 0124, Seville
  - Local Institution - 0123, Valencia
- Turkey (Türkiye) (7):
  - Local Institution - 0107, Ankara
  - Local Institution - 0139, Ankara
  - Local Institution - 0094, Ankara
  - Local Institution - 0096, Antalya
  - Local Institution - 0097, Denizli
  - Local Institution - 0095, Edirne
  - Local Institution - 0146, Istanbul
- United Kingdom (3):
  - Local Institution - 0111, London
  - Local Institution - 0109, Manchester
  - Local Institution - 0140, Truro

REFERENCES:
- [Derived] Viray H, M Mantia C, Jegede OA, Atkins MB, Rosenblatt L, Choueiri TK, McDermott DF, Regan MM. Partitioned overall survival: comprehensive analysis of survival states over 4 years in CheckMate 9ER comparing first-line nivolumab plus cabozantinib versus sunitinib in advanced renal cell carcinoma. J Immunother Cancer. 2026 Jan 30;14(1):e013546. doi: 10.1136/jitc-2025-013546. PMID 41617395
- [Derived] Grimm MO, Karim E, Kapetanakis V, Lothgren M, Ogareva A, Shukla P, Truscott J, Porta C. Two-Stage Estimation of Overall Survival in the Phase 3 CheckMate 9ER Trial, Adjusting for the Impact of Subsequent Therapy. Oncol Ther. 2025 Nov 15. doi: 10.1007/s40487-025-00393-9. Online ahead of print. PMID 41239083
- [Derived] Cella D, Motzer RJ, Suarez C, Blum SI, Ejzykowicz F, Hamilton M, Wallace JF, Simsek B, Zhang J, Ivanescu C, Choueiri TK, Apolo AB. Plain language summary of quality of life in CheckMate 9ER: Cabozantinib plus nivolumab in advanced renal cell carcinoma. Future Oncol. 2025 Jan;21(2):181-194. doi: 10.1080/14796694.2024.2415786. Epub 2024 Oct 25. PMID 39452894
- [Derived] Powles T, Burotto M, Escudier B, Apolo AB, Bourlon MT, Shah AY, Suarez C, Porta C, Barrios CH, Richardet M, Gurney H, Kessler ER, Tomita Y, Bedke J, George S, Scheffold C, Wang P, Fedorov V, Motzer RJ, Choueiri TK. Nivolumab plus cabozantinib versus sunitinib for first-line treatment of advanced renal cell carcinoma: extended follow-up from the phase III randomised CheckMate 9ER trial. ESMO Open. 2024 May;9(5):102994. doi: 10.1016/j.esmoop.2024.102994. Epub 2024 Apr 20. PMID 38642472
- [Derived] Petersohn S, McGregor B, Klijn SL, May JR, Ejzykowicz F, Kurt M, Dyer M, Malcolm B, Branchoux S, Nickel K, George S, Kroep S. Challenges in conducting fractional polynomial and standard parametric network meta-analyses of immune checkpoint inhibitors for first-line advanced renal cell carcinoma. J Comp Eff Res. 2023 Aug;12(8):e230004. doi: 10.57264/cer-2023-0004. Epub 2023 Jul 11. PMID 37431849
- [Derived] Aldin A, Besiroglu B, Adams A, Monsef I, Piechotta V, Tomlinson E, Hornbach C, Dressen N, Goldkuhle M, Maisch P, Dahm P, Heidenreich A, Skoetz N. First-line therapy for adults with advanced renal cell carcinoma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 May 4;5(5):CD013798. doi: 10.1002/14651858.CD013798.pub2. PMID 37146227
- [Derived] Tran BD, Li J, Ly N, Faggioni R, Roskos L. Cabozantinib exposure-response analysis for the phase 3 CheckMate 9ER trial of nivolumab plus cabozantinib versus sunitinib in first-line advanced renal cell carcinoma. Cancer Chemother Pharmacol. 2023 Feb;91(2):179-189. doi: 10.1007/s00280-022-04500-9. Epub 2023 Jan 10. PMID 36625894
- [Derived] Apolo AB, Powles T, Escudier B, Burotto M, Zhang J, Simsek B, Scheffold C, Motzer RJ, Choueiri TK. Nivolumab plus ipilimumab plus cabozantinib triplet combination for patients with previously untreated advanced renal cell carcinoma: Results from a discontinued arm of the phase III CheckMate 9ER trial. Eur J Cancer. 2022 Dec;177:63-71. doi: 10.1016/j.ejca.2022.09.020. Epub 2022 Oct 4. PMID 36327527
- [Derived] Motzer RJ, Powles T, Burotto M, Escudier B, Bourlon MT, Shah AY, Suarez C, Hamzaj A, Porta C, Hocking CM, Kessler ER, Gurney H, Tomita Y, Bedke J, Zhang J, Simsek B, Scheffold C, Apolo AB, Choueiri TK. Nivolumab plus cabozantinib versus sunitinib in first-line treatment for advanced renal cell carcinoma (CheckMate 9ER): long-term follow-up results from an open-label, randomised, phase 3 trial. Lancet Oncol. 2022 Jul;23(7):888-898. doi: 10.1016/S1470-2045(22)00290-X. Epub 2022 Jun 7. PMID 35688173
- [Derived] Cella D, Motzer RJ, Suarez C, Blum SI, Ejzykowicz F, Hamilton M, Wallace JF, Simsek B, Zhang J, Ivanescu C, Apolo AB, Choueiri TK. Patient-reported outcomes with first-line nivolumab plus cabozantinib versus sunitinib in patients with advanced renal cell carcinoma treated in CheckMate 9ER: an open-label, randomised, phase 3 trial. Lancet Oncol. 2022 Feb;23(2):292-303. doi: 10.1016/S1470-2045(21)00693-8. Epub 2022 Jan 12. PMID 35032437
- [Derived] Hamuro L, Hu Z, Passarell J, Barcomb H, Zhang J, Goldstein S, Bello A, Roy A, Zhu L. Exposure-Response Analysis to Support Nivolumab Once Every 4 Weeks Dosing in Combination with Cabozantinib in Renal Cell Carcinoma. Clin Cancer Res. 2022 Apr 14;28(8):1603-1613. doi: 10.1158/1078-0432.CCR-21-3149. PMID 34980597
- [Derived] Choueiri TK, Powles T, Burotto M, Escudier B, Bourlon MT, Zurawski B, Oyervides Juarez VM, Hsieh JJ, Basso U, Shah AY, Suarez C, Hamzaj A, Goh JC, Barrios C, Richardet M, Porta C, Kowalyszyn R, Feregrino JP, Zolnierek J, Pook D, Kessler ER, Tomita Y, Mizuno R, Bedke J, Zhang J, Maurer MA, Simsek B, Ejzykowicz F, Schwab GM, Apolo AB, Motzer RJ; CheckMate 9ER Investigators. Nivolumab plus Cabozantinib versus Sunitinib for Advanced Renal-Cell Carcinoma. N Engl J Med. 2021 Mar 4;384(9):829-841. doi: 10.1056/NEJMoa2026982. PMID 33657295
- [Derived] Hofmann F, Hwang EC, Lam TB, Bex A, Yuan Y, Marconi LS, Ljungberg B. Targeted therapy for metastatic renal cell carcinoma. Cochrane Database Syst Rev. 2020 Oct 14;10(10):CD012796. doi: 10.1002/14651858.CD012796.pub2. PMID 33058158
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT03141177.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 701 participants randomized and 690 treated.
Groups:
- Treatment A: Nivolumab 240 mg flat dose IV Q2W + Cabozantinib 40 mg PO QD
- Treatment B: Nivolumab 3 mg/kg IV Q3W (x4 doses) + Cabozantinib 40 mg PO QD + Ipilimumab 1 mg/kg IV Q3W (x4 doses)
  Then
  Nivolumab 240 mg flat dose IV Q2W + Cabozantinib 40 mg PO QD
- Treatment C: Sunitinib 50 mg PO QD for 4 weeks, followed by 2 weeks off, per cycle
Period: Overall Study
Arm/Group | Treatment A | Treatment B | Treatment C
Started (Started=Randomized) | 323 | 50 | 328
Treated (Treated=Started treatment period) | 320 | 50 | 320
Completed (Completed=Continuing in the Study) | 242 | 34 | 210
Not Completed | 81 | 16 | 118
Not completed — Death | 62 | 13 | 84
Not completed — Participant withdrew consent | 9 | 2 | 13
Not completed — Not reported | 1 | 0 | 1
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Other reasons | 4 | 0 | 11
Not completed — Participants did not start treatment period | 3 | 0 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment A | Treatment B | Treatment C | Total
Number analyzed (Participants) | 323 | 50 | 328 | 701
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.4 (10.2) | 60.3 (9.5) | 60.4 (10.6) | 60.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 16 | 96 | 186
  Male | 249 | 34 | 232 | 515
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 13 | 39 | 90
  Not Hispanic or Latino | 149 | 19 | 151 | 319
  Unknown or Not Reported | 136 | 18 | 138 | 292
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 2 | 5
  Asian | 26 | 0 | 25 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 4 | 5
  White | 267 | 43 | 266 | 576
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 26 | 7 | 31 | 64

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from date of randomization to the first documented tumor progression date or death due to any cause, whichever occurs first based on BICR assessment using RECIST v1.1. Participants who die without a reported progression will be considered to have progressed on the date of their death. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment on or prior to initiation of subsequent anti-cancer therapy. Progressive disease (PD); 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study
Time Frame: From randomization date to date of first documented tumor progression or death, whichever occurs first (Up to 31 months)
Population: All Randomized Participants of treatment A and treatment C
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment C
Number analyzed (Participants) | 323 | 328
Months | 16.59 [12.45 to 24.94] | 8.31 [6.97 to 9.69]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority — Treatment A over Treatment C; p < 0.0001, Stratified Log-Rank; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.41 to 0.64]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time between the date of randomization and the date of death due to any cause. For participants that are alive, their survival time will be censored at the date of last contact date (or "last known alive date").
Time Frame: From randomization date to death date (Up to 31 months)
Population: All Randomized Participants of treatment A and treatment C
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment A | Treatment C
Number analyzed (Participants) | 323 | 328
Months | NA [NA to NA] — Insufficient number of participants with events. | NA [22.6 to NA] — Insufficient number of participants with events.
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority — Treatment A over Treatment C; p = 0.0010, Stratified Log-Rank; Hazard Ratio (HR) = 0.60, 98.89% CI 2-sided [0.40 to 0.89]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the percentage of randomized participants who achieve a best response of confirmed complete response (CR) or confirmed partial response (PR) based on BICR assessments (using RECIST v1.1 criteria) divided by the number of all randomized participants.
  Complete response (CR): Disappearance of all target lesions. Partial response (PR): 30% decrease in the sum of diameters of target lesions.
Time Frame: Up to 31 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 323 | 50 | 328
Percentage of Participants | 55.7 [50.1 to 61.2] | 44.0 [30.0 to 58.7] | 27.1 [22.4 to 32.3]
Statistical Analysis 1: Comparison: Treatment A vs Treatment C; Test type: Superiority — Treatment A over Treatment C; p < 0.0001, Stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 3.52, 95% CI 2-sided [2.51 to 4.95]
Statistical Analysis 2: Comparison: Treatment A vs Treatment C; Test type: Other — Treatment A - Treatment C; Difference of Objective Response Rates = 28.6, 95% CI 2-sided [21.7 to 35.6] — Strata adjusted difference in objective response rate (Nivolumab+Cabozantinib - Sunitinib) based on DerSimonian and Laird

4. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: Number of participants experiencing various types of any grade adverse events (AEs) during the specified time frame.
Time Frame: From first dose to 100 days following last dose (Up to 32 Months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 320 | 50 | 320
Participants | 319 | 50 | 317

5. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs)
Description: Number of participants experiencing various types of any grade serious adverse events (SAEs) during the specified time frame.
Time Frame: From first to dose to 100 days following last dose (Up to 32 months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 320 | 50 | 320
Participants | 160 | 28 | 144

6. Secondary Outcome: Number of Participants Experiencing Adverse Events (AEs) Leading to Discontinuation
Description: Number of participants experiencing various types of any grade adverse events (AEs) leading to discontinuation during the specified time frame.
Time Frame: From first dose to 30 days following last dose (Up to 30 months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 320 | 50 | 320
Participants | 63 | 15 | 54

7. Secondary Outcome: Number of Deaths
Description: Number of deaths due to any cause during the specified time frame.
Time Frame: From first dose to (up to 31 months) following first dose
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 320 | 50 | 320
Participants | 67 | 14 | 99

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Number of participants experiencing laboratory abnormalities in hematology, serum chemistry and electrolytes with grade 3 or higher during the specified time frame.
Time Frame: From first dose to 30 days following last dose (Up to 30 Months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 320 | 50 | 320
Participants
  Hemoglobin: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Hemoglobin: Any grade | 235 | 35 | 256
  Hemoglobin: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Hemoglobin: Grade 3-4 | 9 | 5 | 15
  Platelet Count: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Platelet Count: Any grade | 137 | 27 | 216
  Platelet Count: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Platelet Count: Grade 3-4 | 1 | 0 | 30
  Leukocytes: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Leukocytes: Any grade | 121 | 26 | 207
  Leukocytes: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Leukocytes: Grade 3-4 | 1 | 0 | 16
  Lymphocytes: Any grade: number analyzed (Participants) | 231 | 36 | 231
  Lymphocytes: Any grade | 107 | 22 | 118
  Lymphocytes: Grade 3-4: number analyzed (Participants) | 231 | 36 | 231
  Lymphocytes: Grade 3-4 | 16 | 4 | 24
  Neutrophil: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Neutrophil: Any grade | 115 | 22 | 209
  Neutrophil: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Neutrophil: Grade 3-4 | 10 | 2 | 36
  Alkaline Phosphatase: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Alkaline Phosphatase: Any grade | 194 | 35 | 167
  Alkaline Phosphatase: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Alkaline Phosphatase: Grade 3-4 | 12 | 6 | 6
  Aspartate Aminotransferase (AST): Any grade: number analyzed (Participants) | 317 | 49 | 311
  Aspartate Aminotransferase (AST): Any grade | 260 | 43 | 235
  Aspartate Aminotransferase (AST): Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Aspartate Aminotransferase (AST): Grade 3-4 | 25 | 19 | 8
  Alanine Aminotransferase (ALT): Any grade: number analyzed (Participants) | 317 | 49 | 311
  Alanine Aminotransferase (ALT): Any grade | 268 | 46 | 133
  Alanine Aminotransferase (ALT): Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Alanine Aminotransferase (ALT): Grade 3-4 | 31 | 24 | 11
  Bilirubin: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Bilirubin: Any grade | 57 | 17 | 72
  Bilirubin: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Bilirubin: Grade 3-4 | 3 | 3 | 3
  Creatinine: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Creatinine: Any grade | 221 | 34 | 211
  Creatinine: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Creatinine: Grade 3-4 | 4 | 0 | 2
  Amylase: Any grade: number analyzed (Participants) | 295 | 46 | 283
  Amylase: Any grade | 48 | 28 | 41
  Amylase: Grade 3-4: number analyzed (Participants) | 295 | 46 | 283
  Amylase: Grade 3-4 | 30 | 10 | 17
  Lipase: Any grade: number analyzed (Participants) | 317 | 48 | 306
  Lipase: Any grade | 36 | 27 | 42
  Lipase: Grade 3-4: number analyzed (Participants) | 317 | 48 | 306
  Lipase: Grade 3-4 | 46 | 20 | 41
  Hypernatremia: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Hypernatremia: Any grade | 33 | 7 | 24
  Hypernatremia: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Hypernatremia: Grade 3-4 | 0 | 0 | 0
  Hyponatremia: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Hyponatremia: Any grade | 160 | 31 | 140
  Hyponatremia: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Hyponatremia: Grade 3-4 | 36 | 9 | 41
  Hyperkalemia: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Hyperkalemia: Any grade | 136 | 27 | 100
  Hyperkalemia: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Hyperkalemia: Grade 3-4 | 16 | 2 | 3
  Hypokalemia: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Hypokalemia: Any grade | 64 | 8 | 37
  Hypokalemia: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Hypokalemia: Grade 3-4 | 11 | 0 | 6
  Hypercalcemia: Any grade: number analyzed (Participants) | 315 | 48 | 310
  Hypercalcemia: Any grade | 40 | 9 | 58
  Hypercalcemia: Grade 3-4: number analyzed (Participants) | 315 | 48 | 310
  Hypercalcemia: Grade 3-4 | 1 | 0 | 4
  Hypocalcemia: Any grade: number analyzed (Participants) | 315 | 48 | 310
  Hypocalcemia: Any grade | 174 | 25 | 77
  Hypocalcemia: Grade 3-4: number analyzed (Participants) | 315 | 48 | 310
  Hypocalcemia: Grade 3-4 | 6 | 2 | 2
  Hypermagnesemia: Any grade: number analyzed (Participants) | 316 | 49 | 309
  Hypermagnesemia: Any grade | 42 | 9 | 29
  Hypermagnesemia: Grade 3-4: number analyzed (Participants) | 316 | 49 | 309
  Hypermagnesemia: Grade 3-4 | 12 | 4 | 7
  Hypomagnesemia: Any grade: number analyzed (Participants) | 316 | 49 | 309
  Hypomagnesemia: Any grade | 155 | 18 | 90
  Hypomagnesemia: Grade 3-4: number analyzed (Participants) | 316 | 49 | 309
  Hypomagnesemia: Grade 3-4 | 4 | 1 | 1
  Hyperphosphatemia: Any grade: number analyzed (Participants) | 316 | 49 | 309
  Hyperphosphatemia: Any grade | 0 | 0 | 0
  Hyperphosphatemia: Grade 3-4: number analyzed (Participants) | 316 | 49 | 309
  Hyperphosphatemia: Grade 3-4 | 0 | 0 | 0
  Hypophosphatemia: Any grade: number analyzed (Participants) | 316 | 49 | 309
  Hypophosphatemia: Any grade | 226 | 34 | 154
  Hypophosphatemia: Grade 3-4: number analyzed (Participants) | 316 | 49 | 309
  Hypophosphatemia: Grade 3-4 | 88 | 12 | 31
  Hyperglycemia: Any grade: number analyzed (Participants) | 203 | 37 | 196
  Hyperglycemia: Any grade | 135 | 29 | 139
  Hyperglycemia: Grade 3-4: number analyzed (Participants) | 203 | 37 | 196
  Hyperglycemia: Grade 3-4 | 8 | 2 | 4
  Hypoglycemia: Any grade: number analyzed (Participants) | 308 | 49 | 295
  Hypoglycemia: Any grade | 72 | 10 | 41
  Hypoglycemia: Grade 3-4: number analyzed (Participants) | 308 | 49 | 295
  Hypoglycemia: Grade 3-4 | 2 | 1 | 1

9. Secondary Outcome: Number of Participants With Laboratory Values Grade Shifting From Baseline
Description: Number of participants experiencing worsening shift from baseline in any grade and grade 3-4 of laboratory values during the specified time frame.
Time Frame: From first dose to 30 days following last dose (Up to 30 Months)
Population: All Treated Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 320 | 50 | 320
Participants
  Hemoglobin: Any grade: number analyzed (Participants) | 316 | 49 | 251
  Hemoglobin: Any grade | 117 | 23 | 190
  Hemoglobin: Grade 3-4: number analyzed (Participants) | 316 | 49 | 251
  Hemoglobin: Grade 3-4 | 8 | 5 | 15
  Platelet Count: Any grade: number analyzed (Participants) | 316 | 48 | 310
  Platelet Count: Any grade | 129 | 24 | 216
  Platelet Count: Grade 3-4: number analyzed (Participants) | 316 | 48 | 310
  Platelet Count: Grade 3-4 | 2 | 0 | 30
  Leukocytes: Any grade: number analyzed (Participants) | 316 | 49 | 311
  Leukocytes: Any grade | 116 | 26 | 206
  Leukocytes: Grade 3-4: number analyzed (Participants) | 316 | 49 | 311
  Leukocytes: Grade 3-4 | 1 | 0 | 16
  Lymphocytes: Any grade: number analyzed (Participants) | 228 | 36 | 225
  Lymphocytes: Any grade | 95 | 20 | 102
  Lymphocytes: Grade 3-4: number analyzed (Participants) | 228 | 36 | 225
  Lymphocytes: Grade 3-4 | 15 | 4 | 23
  Neutrophil: Any grade: number analyzed (Participants) | 316 | 49 | 311
  Neutrophil: Any grade | 112 | 22 | 209
  Neutrophil: Grade 3-4: number analyzed (Participants) | 316 | 49 | 311
  Neutrophil: Grade 3-4 | 10 | 2 | 36
  Alkaline Phosphatase: Any grade: number analyzed (Participants) | 317 | 49 | 310
  Alkaline Phosphatase: Any grade | 131 | 31 | 115
  Alkaline Phosphatase: Grade 3-4: number analyzed (Participants) | 317 | 49 | 310
  Alkaline Phosphatase: Grade 3-4 | 9 | 6 | 5
  Aspartate Aminotransferase (AST): Any grade: number analyzed (Participants) | 317 | 49 | 310
  Aspartate Aminotransferase (AST): Any grade | 245 | 42 | 177
  Aspartate Aminotransferase (AST): Grade 3-4: number analyzed (Participants) | 317 | 49 | 310
  Aspartate Aminotransferase (AST): Grade 3-4 | 25 | 19 | 8
  Alanine Aminotransferase (ALT): Any grade: number analyzed (Participants) | 316 | 49 | 310
  Alanine Aminotransferase (ALT): Any grade | 249 | 43 | 121
  Alanine Aminotransferase (ALT) Grade 3-4: number analyzed (Participants) | 316 | 49 | 310
  Alanine Aminotransferase (ALT) Grade 3-4 | 31 | 24 | 11
  Bilirubin: Any grade: number analyzed (Participants) | 316 | 49 | 309
  Bilirubin: Any grade | 55 | 17 | 68
  Bilirubin: Grade 3-4: number analyzed (Participants) | 316 | 49 | 309
  Bilirubin: Grade 3-4 | 3 | 3 | 3
  Creatinine: Any grade: number analyzed (Participants) | 317 | 49 | 311
  Creatinine: Any grade | 123 | 22 | 132
  Creatinine: Grade 3-4: number analyzed (Participants) | 317 | 49 | 311
  Creatinine: Grade 3-4 | 4 | 0 | 2
  Amylase: Any grade: number analyzed (Participants) | 285 | 46 | 277
  Amylase: Any grade | 117 | 26 | 77
  Amylase: Grade 3-4: number analyzed (Participants) | 285 | 46 | 277
  Amylase: Grade 3-4 | 28 | 10 | 16
  Lipase: Any grade: number analyzed (Participants) | 308 | 47 | 300
  Lipase: Any grade | 127 | 27 | 114
  Lipase: Grade 3-4: number analyzed (Participants) | 308 | 47 | 300
  Lipase: Grade 3-4 | 42 | 20 | 40
  Hypernatremia: Any grade: number analyzed (Participants) | 317 | 49 | 310
  Hypernatremia: Any grade | 33 | 7 | 24
  Hypernatremia: Grade 3-4: number analyzed (Participants) | 317 | 49 | 310
  Hypernatremia: Grade 3-4 | 0 | 0 | 0
  Hyponatremia: Any grade: number analyzed (Participants) | 317 | 49 | 310
  Hyponatremia: Any grade | 136 | 30 | 111
  Hyponatremia: Grade 3-4: number analyzed (Participants) | 317 | 49 | 310
  Hyponatremia: Grade 3-4 | 34 | 8 | 37
  Hyperkalemia: Any grade: number analyzed (Participants) | 317 | 49 | 309
  Hyperkalemia: Any grade | 111 | 25 | 82
  Hyperkalemia: Grade 3-4: number analyzed (Participants) | 317 | 49 | 309
  Hyperkalemia: Grade 3-4 | 15 | 2 | 3
  Hypokalemia: Any grade: number analyzed (Participants) | 317 | 49 | 309
  Hypokalemia: Any grade | 61 | 8 | 35
  Hypokalemia: Grade 3-4: number analyzed (Participants) | 317 | 49 | 309
  Hypokalemia: Grade 3-4 | 10 | 0 | 5
  Hypercalcemia: Any grade: number analyzed (Participants) | 314 | 48 | 309
  Hypercalcemia: Any grade | 30 | 7 | 46
  Hypercalcemia: Grade 3-4: number analyzed (Participants) | 314 | 48 | 309
  Hypercalcemia: Grade 3-4 | 1 | 0 | 3
  Hypocalcemia: Any grade: number analyzed (Participants) | 314 | 48 | 309
  Hypocalcemia: Any grade | 170 | 25 | 73
  Hypocalcemia: Grade 3-4: number analyzed (Participants) | 314 | 48 | 309
  Hypocalcemia: Grade 3-4 | 6 | 2 | 2
  Hypermagnesemia: Any grade: number analyzed (Participants) | 308 | 49 | 304
  Hypermagnesemia: Any grade | 38 | 9 | 26
  Hypermagnesemia: Grade 3-4: number analyzed (Participants) | 308 | 49 | 304
  Hypermagnesemia: Grade 3-4 | 12 | 4 | 7
  Hypomagnesemia: Any grade: number analyzed (Participants) | 308 | 49 | 304
  Hypomagnesemia: Any grade | 146 | 16 | 77
  Hypomagnesemia: Grade 3-4: number analyzed (Participants) | 308 | 49 | 304
  Hypomagnesemia: Grade 3-4 | 4 | 1 | 1
  Hyperphosphatemia: Any grade: number analyzed (Participants) | 307 | 49 | 307
  Hyperphosphatemia: Any grade | 0 | 0 | 0
  Hyperphosphatemia: Grade 3-4: number analyzed (Participants) | 307 | 49 | 307
  Hyperphosphatemia: Grade 3-4 | 0 | 0 | 0
  Hypophosphatemia: Any grade: number analyzed (Participants) | 307 | 49 | 307
  Hypophosphatemia: Any grade | 211 | 33 | 147
  Hypophosphatemia: Grade 3-4: number analyzed (Participants) | 307 | 49 | 307
  Hypophosphatemia: Grade 3-4 | 85 | 12 | 31
  Hyperglycemia: Any grade: number analyzed (Participants) | 170 | 33 | 173
  Hyperglycemia: Any grade | 74 | 17 | 76
  Hyperglycemia: Grade 3-4: number analyzed (Participants) | 170 | 33 | 173
  Hyperglycemia: Grade 3-4 | 6 | 2 | 3
  Hypoglycemia: Any grade: number analyzed (Participants) | 262 | 45 | 270
  Hypoglycemia: Any grade | 67 | 9 | 37
  Hypoglycemia: Grade 3-4: number analyzed (Participants) | 262 | 45 | 270
  Hypoglycemia: Grade 3-4 | 2 | 1 | 1

ADVERSE EVENTS:
Time Frame: All cause mortality: From first visit to up to 31 months following first visit SAEs and AEs: From first dose to 100 days following last dose (up to 32 months)
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 67/320 | 14/50 | 99/320
Serious Adverse Events (participants affected / at risk) | 160/320 | 28/50 | 144/320
Other Adverse Events (participants affected / at risk) | 316/320 | 48/50 | 306/320
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=320) | Treatment B (N=50) | Treatment C (N=320)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 11
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 3
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 3 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0 | 2
Intracardiac thrombus (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 2
Myocarditis (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal haemorrhage (Endocrine disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 6 | 2 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0 | 0
Hypophysitis (Endocrine disorders) | 1 | 0 | 0
Hypothalamo-pituitary disorder (Endocrine disorders) | 2 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Thyroiditis acute (Endocrine disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 0 | 4
Anal fistula (Gastrointestinal disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 2
Colitis microscopic (Gastrointestinal disorders) | 1 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 15 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Intussusception (Gastrointestinal disorders) | 1 | 0 | 0
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 5 | 0 | 2
Asthenia (General disorders) | 2 | 1 | 2
Chills (General disorders) | 1 | 0 | 0
Condition aggravated (General disorders) | 0 | 0 | 1
Death (General disorders) | 1 | 1 | 2
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 0 | 1
General physical health deterioration (General disorders) | 2 | 1 | 1
Hernia (General disorders) | 0 | 0 | 1
Inflammation (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 2
Necrosis (General disorders) | 1 | 0 | 0
Pain (General disorders) | 2 | 0 | 6
Pyrexia (General disorders) | 4 | 0 | 5
Sudden death (General disorders) | 1 | 0 | 2
Autoimmune hepatitis (Hepatobiliary disorders) | 1 | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 2 | 2 | 0
Hepatotoxicity (Hepatobiliary disorders) | 2 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
Abdominal sepsis (Infections and infestations) | 0 | 0 | 1
Appendicitis perforated (Infections and infestations) | 2 | 0 | 0
Bronchitis pneumococcal (Infections and infestations) | 1 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Encephalitis (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0 | 0
Large intestine infection (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 0
Lung abscess (Infections and infestations) | 2 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1
Pneumocystis jirovecii infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 9 | 4 | 8
Pneumonia necrotising (Infections and infestations) | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 4 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Soft tissue infection (Infections and infestations) | 2 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 7 | 0 | 5
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radiation injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Bordetella test positive (Investigations) | 1 | 0 | 0
Ejection fraction decreased (Investigations) | 1 | 0 | 1
Escherichia test positive (Investigations) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Human rhinovirus test positive (Investigations) | 1 | 0 | 0
Influenza A virus test positive (Investigations) | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 2
Transaminases increased (Investigations) | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 7 | 1 | 5
Metabolic disorder (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 4
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 24 | 4 | 23
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 4
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 0 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 1
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 2
Seizure (Nervous system disorders) | 2 | 0 | 2
Syncope (Nervous system disorders) | 2 | 2 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 6
Azotaemia (Renal and urinary disorders) | 0 | 0 | 1
Bladder tamponade (Renal and urinary disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 3
Nephritis (Renal and urinary disorders) | 1 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Mediastinal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 1
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 0 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 9
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Peau d'orange (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pemphigoid (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Central venous catheterisation (Surgical and medical procedures) | 0 | 1 | 0
Surgery (Surgical and medical procedures) | 1 | 0 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0 | 0
Bleeding varicose vein (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 1
Embolism (Vascular disorders) | 2 | 0 | 1
Hypertension (Vascular disorders) | 3 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 3
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0 | 1
Vascular occlusion (Vascular disorders) | 1 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment A (N=320) | Treatment B (N=50) | Treatment C (N=320)
Anaemia (Blood and lymphatic system disorders) | 48 | 8 | 85
Leukopenia (Blood and lymphatic system disorders) | 7 | 0 | 24
Neutropenia (Blood and lymphatic system disorders) | 15 | 4 | 50
Thrombocytopenia (Blood and lymphatic system disorders) | 25 | 3 | 62
Hyperthyroidism (Endocrine disorders) | 31 | 3 | 9
Hypothyroidism (Endocrine disorders) | 109 | 15 | 95
Abdominal distension (Gastrointestinal disorders) | 5 | 3 | 7
Abdominal pain (Gastrointestinal disorders) | 50 | 9 | 25
Abdominal pain upper (Gastrointestinal disorders) | 22 | 6 | 21
Colitis (Gastrointestinal disorders) | 6 | 4 | 1
Constipation (Gastrointestinal disorders) | 39 | 12 | 41
Diarrhoea (Gastrointestinal disorders) | 202 | 28 | 151
Dry mouth (Gastrointestinal disorders) | 21 | 3 | 12
Dyspepsia (Gastrointestinal disorders) | 26 | 4 | 40
Gastritis (Gastrointestinal disorders) | 9 | 4 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 25 | 4 | 36
Nausea (Gastrointestinal disorders) | 86 | 15 | 99
Oral dysaesthesia (Gastrointestinal disorders) | 2 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 54 | 8 | 82
Vomiting (Gastrointestinal disorders) | 53 | 10 | 66
Asthenia (General disorders) | 71 | 13 | 58
Chest pain (General disorders) | 8 | 3 | 8
Fatigue (General disorders) | 102 | 19 | 112
Malaise (General disorders) | 12 | 2 | 17
Mucosal inflammation (General disorders) | 66 | 13 | 80
Oedema peripheral (General disorders) | 35 | 8 | 28
Pain (General disorders) | 16 | 4 | 17
Pyrexia (General disorders) | 38 | 12 | 25
Hepatotoxicity (Hepatobiliary disorders) | 16 | 10 | 12
Hypersensitivity (Immune system disorders) | 4 | 3 | 4
Bronchitis (Infections and infestations) | 9 | 3 | 7
Nasopharyngitis (Infections and infestations) | 22 | 5 | 14
Upper respiratory tract infection (Infections and infestations) | 35 | 5 | 12
Urinary tract infection (Infections and infestations) | 23 | 9 | 17
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 3 | 1
Alanine aminotransferase increased (Investigations) | 90 | 21 | 28
Amylase increased (Investigations) | 48 | 8 | 29
Aspartate aminotransferase increased (Investigations) | 82 | 16 | 36
Blood alkaline phosphatase increased (Investigations) | 37 | 8 | 27
Blood bilirubin increased (Investigations) | 18 | 6 | 13
Blood cholesterol increased (Investigations) | 7 | 4 | 10
Blood creatinine increased (Investigations) | 43 | 7 | 43
Blood sodium decreased (Investigations) | 6 | 3 | 2
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 5 | 2
Blood thyroid stimulating hormone increased (Investigations) | 27 | 3 | 20
Lipase increased (Investigations) | 54 | 13 | 38
Lymphocyte count decreased (Investigations) | 6 | 3 | 10
Neutrophil count decreased (Investigations) | 12 | 2 | 27
Platelet count decreased (Investigations) | 18 | 6 | 60
Transaminases increased (Investigations) | 12 | 4 | 5
Weight decreased (Investigations) | 36 | 8 | 10
White blood cell count decreased (Investigations) | 7 | 4 | 18
Decreased appetite (Metabolism and nutrition disorders) | 92 | 15 | 66
Hyperglycaemia (Metabolism and nutrition disorders) | 28 | 3 | 14
Hyperkalaemia (Metabolism and nutrition disorders) | 21 | 4 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 18 | 4 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 22 | 4 | 7
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 3 | 5
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 2 | 11
Hypomagnesaemia (Metabolism and nutrition disorders) | 44 | 3 | 15
Hyponatraemia (Metabolism and nutrition disorders) | 48 | 8 | 28
Hypophosphataemia (Metabolism and nutrition disorders) | 46 | 6 | 18
Arthralgia (Musculoskeletal and connective tissue disorders) | 59 | 7 | 29
Back pain (Musculoskeletal and connective tissue disorders) | 56 | 11 | 38
Muscle spasms (Musculoskeletal and connective tissue disorders) | 38 | 7 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 17 | 3 | 10
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 11 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 | 6 | 29
Dizziness (Nervous system disorders) | 32 | 9 | 19
Dysgeusia (Nervous system disorders) | 76 | 9 | 70
Headache (Nervous system disorders) | 50 | 9 | 36
Paraesthesia (Nervous system disorders) | 11 | 3 | 8
Anxiety (Psychiatric disorders) | 8 | 4 | 9
Depression (Psychiatric disorders) | 15 | 3 | 9
Insomnia (Psychiatric disorders) | 27 | 6 | 17
Proteinuria (Renal and urinary disorders) | 33 | 2 | 25
Renal failure (Renal and urinary disorders) | 10 | 3 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 58 | 14 | 51
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 56 | 7 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 6 | 27
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 2 | 32
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 30 | 5 | 11
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 | 3 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 17 | 3 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 21 | 2 | 15
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 128 | 20 | 130
Pruritus (Skin and subcutaneous tissue disorders) | 60 | 11 | 15
Rash (Skin and subcutaneous tissue disorders) | 69 | 15 | 26
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 27 | 5 | 6
Yellow skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 22
Hypertension (Vascular disorders) | 112 | 18 | 121
Hypotension (Vascular disorders) | 13 | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/77/NCT03141177/Prot_002.pdf
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/77/NCT03141177/SAP_003.pdf